CLINICAL TRIAL: NCT02746835
Title: Physical Condition and Self-efficacy in People With Fall Risk - a Preliminary Study
Brief Title: Physical Condition and Self-efficacy in People With Fall Risk
Acronym: Fall Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Collaborators: Centro de Saúde de Anadia (Unknown)
Responsible Party: Principal Investigator, Marlene Rosa, PhD, Aveiro University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Falls Prevention Program
Record Dates: First submitted 2016-04-11; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Fall Risk
Keywords: physical condition; self-efficacy; fall risk; exercise program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise Protocol (Experimental): Set of exercises for balance, endurance, muscle strength and flexibility
  Interventions: Other: Exercise program for fall prevention

INTERVENTIONS:
Other: Exercise program for fall prevention — Set of exercises to improve the following parameters:
  balance, endurance, muscle strength, flexibility.

SUMMARY:
Middle-aged or older people with fall risk were assessed and invited to a multidisciplinary falls prevention program. This program consisted on an adapted exercise program.

Two sessions per week were performed, during 6 weeks supervised by a physiotherapist.

At the end of this program, measures of physical condition and of self-efficacy were repeated to determine its related-effect.

ELIGIBILITY:
Inclusion Criteria:

* Fall Risk (Morse scale)

Exclusion Criteria:

* Had no capacity to walk independently

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Self-efficacy moving indoors | 6-weeks
  Question 1- Self-efficacy moving indoors; (scoring: 0-not confident - 2-very confident)
Self-efficacy moving outside | 6-weeks
  Question 2 - Self-efficacy moving outside (scoring: 0-not confident - 2-very confident)
Self-efficacy walking uneven surfaces | 6-weeks
  Question 3- Self-efficacy walking through uneven surfaces (scoring: 0-not confident - 2-very confident)
Self-efficacy in physical activities | 6-weeks
  Question 4 - Self-efficacy participating in physical activities (scoring: 0-not confident - 2-very confident)

OTHER OUTCOMES:
Physical Condition related with mobility | 6-weeks
  mobility (5 meters walking test at comfortable speed - 5mWT) (meters/second)
Physical Condition related with balance | 6-weeks
  balance (Functional Reach Test - FRT) (cm)
Physical Condition related with endurance | 6-weeks
  endurance (Sit-to-stand test - STS) (seconds)

CONTACTS AND LOCATIONS:
Locations (1):
- Marlene Cristina Neves Rosa, Anadia, Aveiro District, Portugal